CLINICAL TRIAL: NCT04364893
Title: Suspension of Angiotensin Receptor Blockers and Angiotensin-converting Enzyme Inhibitors and Adverse Outcomes in Hospitalized Patients With Coronavirus Infection (COVID-19). A Randomized Trial
Brief Title: Angiotensin Receptor Blockers and Angiotensin-converting Enzyme Inhibitors and Adverse Outcomes in Patients With COVID19
Acronym: BRACE-CORONA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Brazilian Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRJ_2003
Record Dates: First submitted 2020-04-07; First posted 2020-04-28 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Corona Virus Infection; COVID-19
Keywords: Blockers of angiotensin receptor; Angiotensin-converting enzyme inhibitors; SARS-CoV2
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Suspensions; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Maintenance of Angiotensin Receptor Blockers and Angiotensin-converting Enzyme Inhibitors
  Interventions: Other: Suspension or Maintenance of Angiotensin Receptor Blockers and Angiotensin-converting Enzyme Inhibitors
- Group 2 (Other): Suspension of Angiotensin Receptor Blockers and Angiotensin-converting Enzyme Inhibitors
  Interventions: Other: Suspension or Maintenance of Angiotensin Receptor Blockers and Angiotensin-converting Enzyme Inhibitors

INTERVENTIONS:
Other: Suspension or Maintenance of Angiotensin Receptor Blockers and Angiotensin-converting Enzyme Inhibitors — Suspension or Maintenance of Angiotensin Receptor Blockers and Angiotensin-converting Enzyme Inhibitors

SUMMARY:
Suspension of Angiotensin Receptor Blockers and Angiotensin-converting Enzyme Inhibitors and Adverse Outcomes in Hospitalized Patients With Coronavirus Infection.

DETAILED DESCRIPTION:
Several interactions by pre-existing therapies for chronic diseases, therapies used by SARS-CoV2 infection generate doubts about risks and benefits. Among these situations in which the current data indicate a situation of equipoise would be about the maintenance or suspension of ACEI / BRA in patients with SARS-CoV2 infection. Increasing the expression of ECA-2 could increase the binding to the virus, however, there are studies that indicate this increase in ECA-2 could be protective. So far, there is no clinical evidence to confirm any of the theories, and this question can only be clarified through a randomized clinical trial.

The objective is to evaluate the impact of the suspension of the use of angiotensin-converting enzyme (ACE) inhibitors and angiotensin receptor blockers (BRA) on the length of hospital stay and on the mortality of patients with SARS-CoV2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized with COVID-19 diagnosis using ACE inhibitors or blockers of angiotensin receptor;
* Patients ≥ 18 years old;
* Maximum use of 3 antihypertensive drugs;
* Sign the consent form.

Exclusion Criteria:

* Severe evolution with orotracheal intubation, use of mechanical ventilation and / or hemodynamic instability in the first 24 hours until COVID-19 diagnosis confirmation;
* Patients hospitalized per decompensated congestive heart failure in the last 12 months;
* Use of Sacubitril/Valsartan
* Pregnancy
* Recent acute renal failure and shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2020-04-09 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Median days alive and out of the hospital | 30 days
  The primary outcome of the study will be days alive and outside the hospital (DAOH) at 30 days. This endpoint will be calculated for each included patient and the calculation will be from the date of randomization to the 30-day post-randomization. The DAOH endpoint represents the follow-up time (30 days) subtracted from the hospitalization days and/or the days between death and the end of follow-up.

SECONDARY OUTCOMES:
Number of participants with adverse cardiovascular outcomes and new worsening heart failure | 30 days
  Cardiovascular outcomes such as progression of COVID-19, mortality (general and cardiovascular), acute myocardial infarction, stroke / TIA, new heart failure or worsening of pre-existing HF, myocarditis, pericarditis, arrhythmias requiring treatment, phenomena thromboembolic events, hypertensive crisis, respiratory failure, hemodynamic decompensation, sepsis, renal failure. All events will be reported according to CTCAE 4.0
Cardiovascular biomarkers related to COVID-19 | up to 30 days
  Evaluate levels of biomarkers [troponin, type B natriuretic peptide (BNP), N-terminal natriuretic peptide type B (NT-ProBNP), D-dimer, total lymphocytes , CD4, CD8, macrophages, cytokines, in addition to biomarkers detected by proteomics and metabolomics].

CONTACTS AND LOCATIONS:
Overall Officials: Renato D. Lopes, MD, PhD, Principal Investigator — D'Or Institute for Research and Education
Locations (1):
- Idor, São Paulo, Brazil

REFERENCES:
- [Derived] Macedo AVS, de Barros E Silva PGM, de Paula TC, Moll-Bernardes RJ, Mendonca Dos Santos T, Mazza L, Feldman A, Arruda GDAS, de Albuquerque DC, de Sousa AS, de Souza OF, Gibson CM, Granger CB, Alexander JH, Lopes RD. Discontinuing vs continuing ACEIs and ARBs in hospitalized patients with COVID-19 according to disease severity: Insights from the BRACE CORONA trial. Am Heart J. 2022 Jul;249:86-97. doi: 10.1016/j.ahj.2022.04.001. Epub 2022 Apr 8. PMID 35405099
- [Derived] Lopes RD, Macedo AVS, de Barros E Silva PGM, Moll-Bernardes RJ, Dos Santos TM, Mazza L, Feldman A, D'Andrea Saba Arruda G, de Albuquerque DC, Camiletti AS, de Sousa AS, de Paula TC, Giusti KGD, Domiciano RAM, Noya-Rabelo MM, Hamilton AM, Loures VA, Dionisio RM, Furquim TAB, De Luca FA, Dos Santos Sousa IB, Bandeira BS, Zukowski CN, de Oliveira RGG, Ribeiro NB, de Moraes JL, Petriz JLF, Pimentel AM, Miranda JS, de Jesus Abufaiad BE, Gibson CM, Granger CB, Alexander JH, de Souza OF; BRACE CORONA Investigators. Effect of Discontinuing vs Continuing Angiotensin-Converting Enzyme Inhibitors and Angiotensin II Receptor Blockers on Days Alive and Out of the Hospital in Patients Admitted With COVID-19: A Randomized Clinical Trial. JAMA. 2021 Jan 19;325(3):254-264. doi: 10.1001/jama.2020.25864. PMID 33464336